CLINICAL TRIAL: NCT01564667
Title: Attention Bias Modification Treatment for Warzone-Related PTSD: A Randomized Clinical Trial Magnetoencephalography Study
Brief Title: Attention Bias Modification Treatment for Warzone-Related Posttraumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: At Ease USA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-16311
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; Posttraumatic Stress; Post Traumatic Stress; Attention Bias; Threat Bias; Combat; Warzone
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Attention Bias Modification Treatment (Experimental): Attention bias modification training using a computerized spatial attention task (dot-probe) designed to alter threat-bias attention patterns away from threat.
  Interventions: Behavioral: Attention Bias Modification Training Protocol
- Attentional Control Training (Active Comparator): Attention control training using a computerized spatial attention taks (dot-probe) counter balances training toward and away from threat.
  Interventions: Behavioral: Attention Bias Modification Training Protocol

INTERVENTIONS:
Behavioral: Attention Bias Modification Training Protocol — Attention Bias Modification computerized training sessions administered 2 times per week for 4 weeks making a total of 8 training sessions.

SUMMARY:
Veterans with Posttraumatic Stress Disorder (PTSD) will be randomly assigned to either Attention Bias Modification Treatment (ABMT) designed to reduce bias toward threat or a placebo control condition not designed to change attention patterns. Outcome measures will be PTSD, anxiety, depression, and alexithymia symptoms as measured by standard psychological interviews and questionnaires. Participants will also be invited to participate in physiological testing before and after receiving AMBT or placebo to serve as additional outcome measures and assess brain functioning, heart rate, and muscle tension.

The investigators expect to see significant PTSD symptom reduction in the Attention Bias Modification Treatment (ABMT) group relative to the placebo control group in which no symptomatic relief is expected. At the end of the study, if ABMT is shown to be effective, we will offer active ABMT to those participants randomly assigned to the placebo arm if they would like to receive the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with Posttraumatic Stress Disorder (PTSD) serving in United States Military after March 20, 2003.

Exclusion Criteria:

* Schizophrenia
* Bipolar Disorder
* Obsessive Compulsive Disorder
* Head Injury with Loss of Consciousness for more than 30 minutes
* Active Alcohol/Substance Dependence in past 6 months

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Will Posttraumatic Stress Disorder and Symptom decrease with intervention | 8 weeks
  Using Clinician-Administered PTSD Scale (CAPS): The clinician-Administered PTSD Scale (CAPS) is a 30-item structured interview that corresponds to the DSM-IV criteria for PTSD (Blake, Weathers, Nagy, Kaloupek, Charney, & Keane, 1995) to assess symptoms of PTSD outcome.

SECONDARY OUTCOMES:
Other psychiatics symptoms (ie Depression, Anger, Anxiety) | 8 weeks
  To assess potential decrease in psychiatric symptoms associated with PTSD, by comparing pre intervention and post intervention scores on psychological measures of deprssion, anger and anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Amy S Badura Brack, PhD, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States

REFERENCES:
- [Background] Hakamata Y, Lissek S, Bar-Haim Y, Britton JC, Fox NA, Leibenluft E, Ernst M, Pine DS. Attention bias modification treatment: a meta-analysis toward the establishment of novel treatment for anxiety. Biol Psychiatry. 2010 Dec 1;68(11):982-90. doi: 10.1016/j.biopsych.2010.07.021. PMID 20887977
- [Derived] Badura-Brack AS, Naim R, Ryan TJ, Levy O, Abend R, Khanna MM, McDermott TJ, Pine DS, Bar-Haim Y. Effect of Attention Training on Attention Bias Variability and PTSD Symptoms: Randomized Controlled Trials in Israeli and U.S. Combat Veterans. Am J Psychiatry. 2015 Dec;172(12):1233-41. doi: 10.1176/appi.ajp.2015.14121578. Epub 2015 Jul 24. PMID 26206075